CLINICAL TRIAL: NCT03431454
Title: Comparison of Three Vision Therapy Approaches for Convergence Insufficiency
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Shahid Beheshti University of Medical Sciences, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 92149
Record Dates: First submitted 2017-12-12; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2017-12

CONDITIONS: Comparison of Three Vision Therapy Approaches for Convergence Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- home-based vision orthoptic therapy (HBVOT) group (Active Comparator): In the home-based vision orthoptic therapy (HBVOT) group, patients were trained to do the pencil push-ups procedure 15 minutes per day, five days a week
  Interventions: Procedure: trained to do the pencil push-ups procedure
- office-based vision orthoptic therapy (OBVOT) group (Active Comparator): In the office-based vision orthoptic therapy (OBVOT) group, 60 minutes of orthoptic therapy using a major amblyoscope twice weekly with additional home orthoptic therapy was prescribed
  Interventions: Procedure: using a major amblyoscope twice weekly with additional home orthoptic therapy
- augmented office-based vision orthoptic therapy (AOBVOT) group (Active Comparator): For the augmented office-based vision orthoptic therapy (AOBVOT) group, orthoptic exercises using three diopter over-minus lenses and a base out prism, in addition to major amblyoscope and additional home reinforcement was prescribed in the same period of time.
  Interventions: Procedure: using three diopter over-minus lenses and a base out prism

INTERVENTIONS:
Procedure: trained to do the pencil push-ups procedure — 15 minutes per day, five days a week
  Arms: home-based vision orthoptic therapy (HBVOT) group
Procedure: using a major amblyoscope twice weekly with additional home orthoptic therapy — 60 minutes of orthoptic therapy using a major amblyoscope twice weekly with additional home orthoptic therapy was prescribed.
  Arms: office-based vision orthoptic therapy (OBVOT) group
Procedure: using three diopter over-minus lenses and a base out prism — For the augmented office-based vision orthoptic therapy (AOBVOT) group, orthoptic exercises using three diopter over-minus lenses and a base out prism, in addition to major amblyoscope and additional home reinforcement was prescribed in the same period of time.
  Arms: augmented office-based vision orthoptic therapy (AOBVOT) group

SUMMARY:
We compared the effectiveness of three active vision therapy approaches for convergence insufficiency (CI). Patients with eligible criteria and symptomatic CI were included in a prospective study and randomly allocated into three groups. In the home-based vision orthoptic therapy (HBVOT) group, patients were trained to do the pencil push-ups procedure 15 minutes per day, five days a week. In the office-based vision orthoptic therapy (OBVOT) group, 60 minutes of orthoptic therapy using a major amblyoscope twice weekly with additional home orthoptic therapy was prescribed. For the augmented office-based vision orthoptic therapy (AOBVOT) group, orthoptic exercises using three diopter over-minus lenses and a base out prism, in addition to major amblyoscope and additional home reinforcement was prescribed in the same period of time.

ELIGIBILITY:
Inclusion Criteria:

* patients between 15 and 35 years of age who have symptomatic CI using the Convergence Insufficiency Symptom Survey (CISS) scoring system.
* best-corrected visual acuity ≥ 20/25
* exophoria at near at least 4 prism diopters (△) greater than at distance
* near point of convergence more than 6.0 cm break
* insufficient positive fusional vergence (PFV) (failing Sheard's criterion or PFV ≤ 15 △ base-out) at near distance.

Exclusion Criteria:

* amblyopia (VA worse than 20/30 in each eye), presence of manifest strabismus, history of ocular surgery, any systemic disorder, anisometropia of more than 1.5 diopter of myopia or hyperopia or significant refractive error, and nystagmus and usage of medications that may impair accommodation or convergence. ,ocular surface abnormalities or history of ocular allergy or those who had previously been treated for CI

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
symptomatic convergence insufficiency | one month
  A symptomatic score was an average score of 16 or higher on the CISS(conv-insuff-sympt-scove)

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran

REFERENCES:
- [Derived] Scheiman M, Kulp MT, Cotter SA, Lawrenson JG, Wang L, Li T. Interventions for convergence insufficiency: a network meta-analysis. Cochrane Database Syst Rev. 2020 Dec 2;12(12):CD006768. doi: 10.1002/14651858.CD006768.pub3. PMID 33263359